CLINICAL TRIAL: NCT03338153
Title: Evaluation of Long-term Coronary Stenting Outcomes in Diabetic Patients With or Without Optimal Glycemic Control Referring to Tehran Heart Center Since June 2007 to June 2009
Brief Title: Evaluation of Long-term Coronary Stenting Outcomes in Diabetic Patients With or Without Optimal Glycemic Control
Status: Completed | Type: Observational
Sponsor: Tehran Heart Center (Other)
Responsible Party: Sponsor
Other Study IDs: TUMS-90-04-30-15887
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Diabetes; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- controlled diabetes: diabetic patients with HbA1C level below 7.0%
- uncontrolled diabetes: diabetic patients with hbA1C level above 7%
- non-diabetic: patients who does not have diabetes at the time of PCI

SUMMARY:
the purpose of this study is to determine whether appropriate control of diabetes around the PCI time is related with MACE and outcome of diabetic patients.

DETAILED DESCRIPTION:
Despite recent advances in coronary revascularization, cardiovascular disease accounts for about 75% of all hospital admissions in diabetic patients.although the introduction of drug-eluting stents has reduced the rates of restenosis after PCI, diabetic patients undergoing PCI will have poorer clinical outcomes.In this study, we sought to investigate whether a pre and post procedural glycemic control in diabetic patients,as reflected by HgbA1C prior,1 and 6 months after elective PCI,was related to major advance cardiac events (MACE) during 3 year follow up.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-75
* coronary stenosis > 70%

Exclusion Criteria:

* Myocardial infarction in 72 hours prior to PCI
* LVEF < 30%
* Residual Stenosis>30%
* Cr level > 2.0
* hemodynamic compromise during intervention
* Left main lesions
* PCI for vein grafts

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing per-cutaneous coronary intervention between October 2007 and December 2009
Sampling Method: Probability Sample
Enrollment: 1353 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac event | during 3 years after per-cutaneous coronary intervention

SECONDARY OUTCOMES:
target vessel revascularization | during 3 years after PCI
target lesion revascularization | during 3 years after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim kassaian, MD, Principal Investigator — Tehran Heart Center
Locations (1):
- Tehran heart center, Tehran university of medical sciences, Tehran, Iran